CLINICAL TRIAL: NCT00203346
Title: Greater Occipital Nerve (GON) Block for Migraine
Brief Title: Research Study Examining Nerve Block for Migraine
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Other Study IDs: WBY/GON
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Greater Occipital Nerve Block

SUMMARY:
Migraine and the skin sensitivity that accompanies it can go away in minutes after a nerve block, which is a procedure involving an injection of a small amount of a local anesthetic next to a nerve to the skin, causing an area of skin to become numb. We have also noticed that light sensitivity goes away quickly after a nerve block. We would like to see how quickly this happens and how long the benefit of nerve block lasts. We are interested to see if these effects are due to the injection itself or due to the lidocaine.

A subject may be asked to participate in this study if a subjects physician has planned for a subject to receive an injection of BOTOX® in the area of the Greater Occipital Nerve (a spinal nerve located at the back of the head) as part of a subjects routine preventive treatment for migraine today.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with episodic or transformed migraine age 18to 80 years old.
* Subjects must have unilateral migraine headache and trigeminal distribution brush allodynia at the time of injection.
* Subjects must be able to consent or assent to the study.

Exclusion Criteria:

* Subjects who in their own or in the investigator's opinion are unable to report the severity of four symptoms (pin sharpness to determine efficacy of nerve block, headache severity, photophobia severity and allodynia severity), every 30 seconds for 5 minutes post injection;
* Subjects with skull defect, or history of injury to the area of the GON.
* Subjects with prior adverse reaction to GON block, lidocaine or marcaine.
* Subjects who are pregnant or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: William B Young, MD, Principal Investigator — Thomas Jefferson University, Jefferson Headache Center
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States